CLINICAL TRIAL: NCT05029544
Title: Comparison of Effects of Kinesio Taping and Dynamic Taping Added to a Rehabilitation Programme for Patients With Symptomatic Rotator Cuff Tendinopathy: A Randomised Controlled Trial
Brief Title: Dynamic Taping in Symptomatic Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Meltem Koc, Research Asisstant, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: interventional
Record Dates: First submitted 2021-08-19; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Rotator Cuff Tendinosis
Keywords: Rotatory cuff tendinopathy; Acromiohumeral distance; Dynamic taping; Kinesiotaping; Proprioception; Shoulder pain; Rehabilitation
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain | interventions — Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Only the investigator who performed the acromiohumeral distance measurements was blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention group 1 (Active Comparator): dynamic taping and standard rehabilitation program
  Interventions: Other: Dynamic taping; Other: Physiotherapy and Rehabilitation
- intervention group 2 (Active Comparator): Kinesio taping and standard rehabilitation program
  Interventions: Other: Kinesio taping; Other: Physiotherapy and Rehabilitation
- Control group (Other): No taping on shoulder, only standard rehabilitation program
  Interventions: Other: Physiotherapy and Rehabilitation

INTERVENTIONS:
Other: Dynamic taping — The intervention of this experimental study was therapeutic taping (dynamic tape) on the symptomatic shoulders of the participants.
  Arms: intervention group 1
Other: Kinesio taping — The intervention of this experimental study was therapeutic taping (kinesio tape) on the symptomatic shoulders of the participants.
  Arms: intervention group 2
Other: Physiotherapy and Rehabilitation — exercise, manuel therapy, mobilization, massage, sensorimotor control

SUMMARY:
This study was conducted to compare the efficacy of two different therapeutic bands in symptomatic rotator cuff tendinopathy. One of the tapes was kinesio tape and the other was dynamic tape. The study was in a parallel group randomized controlled trial design.

DETAILED DESCRIPTION:
This study was planned to compare the effectiveness of dynamic taping and kinesio taping combined with a rehabilitation program on the symptomatic shoulder in patients with symptomatic rotator cuff tendinopathy (RCT). The study was carried out on 60 patients who applied to Muğla Training and Research Hospital Physical Therapy and Rehabilitation outpatient clinic with symptoms of RCT. The patients were divided into 3 groups by randomization method. Dynamic taping was applied to the symptomatic shoulder in the first group and kinesio taping was performed in the second group. The third group was the control group and no taping was done. A standard rehabilitation program was applied for the individuals in the whole group. Evaluations were made before and after treatment (6 weeks). Evaluation parameters were acromiohumeral distance (primary outcome), shoulder joint range of motion, muscle strength, proprioception measurements, and function evaluations. The acromiohumeral distance was measured by the radiologist, and all other measurements and treatments were performed by the physiotherapist. Standard goniometer was used for shoulder joint range of motion measurement, manual muscle dynamometer was used for muscle strength measurement, and digital inclinometer was used for proprioception measurement. Timed arm-shoulder function test was performed for function evaluation. The arm, shoulder, and hand disability (DASH) questionnaire and the Western Ontario Rotator Cuff Index (WORC) were used for the self-function report. The data obtained from the research will be analyzed using the SPSS program. Statistical significance level will be accepted as p<0.05. In the statistical difference analysis between groups, one-way ANOVA test will be used for parametric data and Kruskal-Wallis test will be used for non-parametric data.

ELIGIBILITY:
Inclusion Criteria:

* Those with a diagnosis of RCT
* Those with subacromial pain
* At least two of the three impingement tests are positive (empty-can test, Hawkins-Kennedy test, modified Neer test)
* 18-65 years old

Exclusion Criteria:

* Those with open wounds at the taping area
* Those who have allergic reactions to taping
* Those who have had shoulder surgery before
* Those with total rotator cuff tendon rupture
* Those with a history of fractures in the upper extremity or glenohumeral joint subluxation -- Presence of adhesive capsulitis (those with more than passive shoulder joint motion loss 70%)
* Presence of congenital or acquired deformity involving the upper extremity
* Those with rheumatic or neurologic disease
* Those with cervical radiculopathy
* Those with a history of neoplasm or cognitive impairment (MMSE<24)
* Those who received corticosteroid injection to the shoulder region in the last 3 months
* Those who received physiotherapy treatment in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Acromiohumeral Distance (AHD) | Change in acromiohumeral distance at 6 week
  Measurement of the distance between the humeral head and the inferior acromion by ultrasound to determine the subacromial space

SECONDARY OUTCOMES:
Proprioception | Change in proprioception at 6 week
  Measurement with digital inclinometer with active reposition repetition method in shoulder flexion of 30 and 60 degrees
Muscle Strength | Change in shoulder muscle strength at 6 week
  shoulder muscle strength measurement (flexion, abduction, internal and external rotation) with a manual dynamometer
Shoulder Range of Motion | Change in shoulder range of motion at 6 week
  Shoulder range of motion (painless and full) measurement (flexion, abduction, internal and external rotation)
Lateral Scapular Slide Test | Change in scapular position at 6 week
  Background: The Lateral Scapular Slide Test is a static test used in clinical settings to assess medio-lateral inferior angle displacement and scapular asymmetry at three different degrees of shoulder abduction.
Timed Functional Arm and Shoulder Test | Change in shoulder function at 6 week
  The test includes 3 steps. 1) Hand to head and back: this test is timed for 30 seconds. Each time the patient touches the back of his or her head, it counts as 1 repetition. 2) Wall wash outward and inward: this test is timed for 60 seconds in each direction. 3) Gallon-jug lift: this test is timed for 30 seconds. Starting counter height should be 36 inches, and the shelf should be 20 inches above the counter (56 inches off the floor). Begin with a full gallon jug on the counter. Lift the jug to touch the shelf and return to start. Every time the jug touches the shelf, it counts as 1 repetition. Record the score.
The Disabilities of the Arm, Shoulder and Hand (DASH) | Change in DASH scores at 6 week
  DASH questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale. In DASH higher scores indicate a greater level of disability and severity, whereas, lower scores indicate a lower level of disability. The score ranges from 0 (no disability) to 100 (most severe disability).
Western Ontario Rotator Cuff (WORC) Index | Change in WORC scores at 6 week
  the WORC Index, is a disease-specific quality of life questionnaire, evaluating the change in symptoms and functional ability, specific to a RC tendinopathy. Each question uses a visual analogue scale (VAS) - which is a straight line, representing a 100-point scale, ranging from 0-100. The maximum score (21items) is 2100 (worst possible symptoms). Zero (0) represents no symptoms at all. To make the final score more clinically friendly, some minor math is involved. The score can be reported as a percentage by subtracting the total from 2100, dividing by 2100, and multiplying by 100. This give an overall percentage. Total final WORC scores can, therefore, range from 0% ( lowest functional status level) to 100% (the highest functional status).

CONTACTS AND LOCATIONS:
Overall Officials: Kılıçhan Bayar, Prof, Study Chair — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Sıtkı Koçman University, Muğla, Turkey (Türkiye)